CLINICAL TRIAL: NCT04080167
Title: Integration of mHEALTH Into the Care of Patients With Sickle Cell Disease to Increase Hydroxyurea Utilization- mESH Study
Brief Title: Integration of mHEALTH Into the Care of Patients With Sickle Cell Disease to Increase Hydroxyurea Utilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: RTI International (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: mESH; 5U01HL133996 (NIH)
Record Dates: First submitted 2019-08-15; First posted 2019-09-06 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Sickle Cell Disease
Keywords: implementation science; sickle cell anemia; digital medicine; adherence; hydroxycarbamide; health innovation
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: nonrandomized, closed cohort, stepped-wedge cluster trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (InCharge Health app) (Other): Patient receives the InCharge Health app for 6 months
  Interventions: Behavioral: InCharge Health mobile application
- Arm 2 (HU Toolbox app) (Other): Provider receives the HU Toolbox app for 9 months
  Interventions: Behavioral: HU Toolbox mobile application

INTERVENTIONS:
Behavioral: InCharge Health mobile application — The InCharge Health app features include: Daily reminders; Ability to customize content of message and time of day when the message comes; Symptom tracker to monitor daily pain and mood; 7-day streak that tracks daily adherence; Graphing adherence against pain symptoms; Communication feature allowing the patient to connect to the clinic and a "health partner"; Link to discussion forum where communication to other patients can occur; Education bank that provides information about SCD and hydroxyurea. Participants can delay daily push notifications. If hospitalized, participants may stop notifications. A special feature of the app is to set up a "health partner", who may be a person the participant may choose from his/her contact list and who will receive notifications if it had been <4 hours since not documenting the use of hydroxyurea. The "app healthy partner" will be encouraged to message the participant to remind him/her to take the medication.
  Arms: Arm 1 (InCharge Health app)
Behavioral: HU Toolbox mobile application — The HU Toolbox app includes algorithms for hydroxyurea use and is ready for immediate use on Apple and Android operating systems. In addition, it has the NHLBI guidelines adapted for pediatrics (guidelines/recommendations separated by age) and for adults (guidelines/ recommendations separated by organ system, laboratory, or physical exam finding). The HU Toolbox app includes the ability to search guidelines for key words and add notes. Algorithms are also included as PDF documents that can be printed out or emailed. Finally, a contact list of local SCD specialists and important contacts is included, so providers can easily contact SCD experts and expect an answer in 24 hours or less. The HU Toolbox app is easily updated with all data and resources stored on a cloud-based server that can provide instant up-to-date information to those using the app.
  Arms: Arm 2 (HU Toolbox app)

SUMMARY:
This project proposes to develop, test and evaluate targeted interventions to improve clinical provider prescribing of and patient adherence to hydroxyurea (HU). Using a stepped-wedge design, The investigators will test two innovative interventions utilizing mobile health to address both patients' and providers' needs: 1) an mHealth application for patients (InCharge Health app) that includes multi-component features to address the memory, motivation, and knowledge barriers to hydroxyurea use, and 2) an mHealth toolbox application for providers (HU Toolbox app) that addresses clinical knowledge barriers in prescribing and monitoring hydroxyurea use. These two interventions will be tested through the following aims:

Aim 1. Improve Patient Adherence to Hydroxyurea: Addressing Memory, Motivation, and Knowledge Barriers to Hydroxyurea Use. Primary hypothesis: The investigators hypothesize that among adolescents and adults with SCD, the adherence to hydroxyurea, as measured by percentage of days covered (PDC), will increase by at least 20% at 24 weeks after receiving the InCharge Health app, compared to their hydroxyurea adherence at baseline.

Sub-aim 1.a. To examine and assess both patient engagement and behaviors related to use of the InCharge Health app, the investigators will evaluate consistent use of the app among enrolled patients, patient satisfaction, and continued use of the app beyond the study period.

Sub-Aim 1.b. To examine the clinical influence of the use of the InCharge Health app on PDC, patients' clinical outcomes, perceived health literacy, health related quality of life, and perceived self-efficacy between baseline and 24 weeks.

Aim 2. Improve Provider Hydroxyurea Awareness, Prescribing and Monitoring Behaviors.

Sub-Aim 2.a. To examine and assess provider engagement and behaviors related to use of the HU Toolbox, the investigators will evaluate consistent use of the app among enrolled providers, providers' satisfaction, and continued use of the app beyond the study period.

Sub-Aim 2.b. To assess the combined effects of the patient and provider mHealth interventions on hydroxyurea and health care utilization, the investigators will examine if the changes in hydroxyurea adherence are enhanced by the use of both provider and patient interventions compared to those not exposed to one or both interventions.

Aim 3. Identify and Evaluate the Barriers and Facilitators to the use of mHealth Interventions.

DETAILED DESCRIPTION:
The National Heart, Lung, and Blood Institute (NHLBI) created the Sickle Cell Disease Implementation Consortium (SCDIC) to apply implementation science methods to identify and address barriers to guideline-based care in sickle cell disease (SCD) and promote evidence-based treatment for SCD patients between ages 15 to 45 years. The SCDIC conducted a systematic literature review and a comprehensive needs assessment among the eight participating centers. A major conclusion was that care redesign to support better hydroxyurea utilization would likely improve clinical outcomes for patients with SCD. Hydroxyurea therapy has been shown to improve patient outcomes and reduce disease complications and is endorsed by the NHLBI. SCDIC now proposes to develop, test and evaluate targeted interventions to improve clinical provider prescribing of and patient adherence to hydroxyurea.

The overall purpose of this proposed project is to address barriers identified by the needs assessment to improve adherence with hydroxyurea therapy. Multiple approaches for improving adherence with pharmaceutical regimens have been studied and demonstrate a need to address barriers that both providers and patients face. This project aims, via a stepped-wedge design, to test two innovative interventions utilizing mobile health (mHealth), to address both patients' and providers' needs: 1) an mHealth application for patients (InCharge Health app) that includes multi-component features to address the memory, motivation, and knowledge barriers to hydroxyurea use, and 2) an mHealth toolbox application for providers (HU Toolbox app) that addresses the clinical knowledge barriers in prescribing and monitoring hydroxyurea use. These two interventions will be tested through the following aims:

Aim 1. Improve Patient Adherence to Hydroxyurea: Addressing Memory, Motivation, and Knowledge Barriers to Hydroxyurea Use. Primary hypothesis: The investigators hypothesize that among adolescents and adults with SCD, the adherence to hydroxyurea, as measured by percentage of days covered (PDC), will increase by at least 20% at 24 weeks after receiving the InCharge Health app, compared to their hydroxyurea adherence at baseline.

Sub-aim 1.a. To examine and assess both patient engagement and behaviors related to use of the InCharge Health app, the investigators will evaluate consistent use of the app among enrolled patients, patient satisfaction, and continued use of the app beyond the study period.

Sub-Aim 1.b. To examine the clinical influence of the use of the InCharge Health app on PDC, patients' clinical outcomes, perceived health literacy, health related quality of life, and perceived self-efficacy between baseline and 24 weeks.

Aim 2. Improve Provider Hydroxyurea Awareness, Prescribing and Monitoring Behaviors. The investigators will examine among providers using the HU Toolbox App if there is an increase in reported awareness of hydroxyurea benefits and risks, accurate prescribing of hydroxyurea, and perceived self-efficacy to correctly administer hydroxyurea therapy between baseline and after 9 months of using the HU Toolbox app.

Sub-Aim 2.a. To examine and assess provider engagement and behaviors related to use of the HU Toolbox, the investigators will evaluate consistent use of the app among enrolled providers, providers' satisfaction, and continued use of the app beyond the study period.

Sub-Aim 2.b. To assess the combined effects of the patient and provider mHealth interventions on hydroxyurea and health care utilization, the investigators will examine if the changes in hydroxyurea adherence are enhanced by the use of both provider and patient interventions compared to those not exposed to one or both interventions.

Aim 3. Identify and Evaluate the Barriers and Facilitators to the use of mHealth Interventions. The investigators will evaluate the strategies used by participating sites in supporting the implementation of mHealth interventions via a mixed-method evaluation of the facilitators and barriers in adopting and implementing the mHealth interventions from multiple stakeholder perspectives: patient, provider, and organization.

Both mHealth interventions will be tested concurrently and because the investigators are using a stepped-wedge design, each site will enter the study at different times. Provider participants will receive the HU Toolbox intervention for 9 months with a lagged but overlapping introduction of the InCharge Health intervention patient participants for 24 weeks. The implementation evaluation will be guided by RE-AIM to assess the Reach, Effectiveness, Adoption, Implementation and Maintenance of the interventions. All sites will also complete follow-on needs assessment and medical record abstractions that will provide data to evaluate other patient and provider outcomes, barriers and enablers to hydroxyurea prescribing, use, and monitoring.

mHealth technology can be leveraged to support more effective use of hydroxyurea and eventually improved SCD clinical outcomes. If the mHealth applications tested in this study show preliminary efficacy, both apps could be scaled up within SCDIC centers and expanded to other institutions outside the SCDIC.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 years up to and including 45 years
* Treated at or affiliated with one of the SCDIC sites
* English speaking
* Confirmed Sickle Cell Disease (SCD) diagnosis. An SCD diagnosis is defined as Hb fractionation test (e.g., high- performance liquid chromatography or another technique) that is diagnostic of one the following: Hb SS, Hb SC, Hb Sβ-thalassemia, Hb SO, Hb SD, Hb SG, Hb SE, or Hb SF.
* Willing and cognitively able to give informed consent
* Access to a cellular/mobile smart phone (either Android or IPhone are acceptable)
* Hydroxyurea therapy: Already receiving hydroxyurea therapy: defined as at least one prior prescription to hydroxyurea in the past 3 months and no plans to escalate the dose by more than 5 mg/kg/day. Initiating hydroxyurea therapy: defined as at least one prescription written at the time of study enrollment (the first prescription must be written on the same day as study enrollment). Patients who initiate hydroxyurea on the same day of study enrollment will not contribute to the total of 46 patients target accrual for the site. A max of 30 patients who are initiating hydroxyurea can be enrolled per site.

Exclusion Criteria:

* Current pregnancy
* On a chronic transfusion program in which they receive more than 8 erythrocyte transfusions in a 12-month period.
* A red blood cell transfusion in the past 60 days
* Currently using another phone application or an online-based tool (e-health tool) to increase hydroxyurea adherence

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 382 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Hankins, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (7):
- United States (7):
  - Georgia Regents University, Augusta, Georgia
  - University of Illinois, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient-level data will be available to researchers outside the SCDIC through an application and approval process through BIOLINCC. To protect the confidentiality and privacy of the participants, investigators granted access to the limited access data must adhere to strict requirements incorporated into a standard Data Use Agreement. In accordance with NHLBI policy, outside researchers may also be required to submit an approval to BIOLINCC from their IRB.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available by BIOLINCC for the study, upon request.
Access Criteria: Access to the data must be requested through BIOLINCC by first creating an account and submitting a request for the data through the BIOLINCC website.
URL: http://biolincc.nhlbi.nih.gov/register

REFERENCES:
- [Background] Badawy SM, DiMartino L, Brambilla D, Klesges L, Baumann A, Burns E, DeMartino T, Jacobs S, Khan H, Nwosu C, Shah N, Hankins JS; Sickle Cell Disease Implementation Consortium. Impact of the COVID-19 Pandemic on the Implementation of Mobile Health to Improve the Uptake of Hydroxyurea in Patients With Sickle Cell Disease: Mixed Methods Study. JMIR Form Res. 2022 Oct 14;6(10):e41415. doi: 10.2196/41415. PMID 36240004
- [Derived] Hankins JS, Brambilla D, Potter MB, Kutlar A, Gibson R, King AA, Baumann AA, Melvin C, Gordeuk VR, Hsu LL, Nwosu C, Porter JS, Alberts NM, Badawy SM, Simon J, Glassberg JA, Lottenberg R, DiMartino L, Jacobs S, Fernandez ME, Bosworth HB, Klesges LM, Shah N. A multilevel mHealth intervention boosts adherence to hydroxyurea in individuals with sickle cell disease. Blood Adv. 2023 Dec 12;7(23):7190-7201. doi: 10.1182/bloodadvances.2023010670. PMID 37738155
- [Derived] Hankins JS, Shah N, DiMartino L, Brambilla D, Fernandez ME, Gibson RW, Gordeuk VR, Lottenberg R, Kutlar A, Melvin C, Simon J, Wun T, Treadwell M, Calhoun C, Baumann A, Potter MB, Klesges L, Bosworth H; Sickle Cell Disease Implementation Consortium. Integration of Mobile Health Into Sickle Cell Disease Care to Increase Hydroxyurea Utilization: Protocol for an Efficacy and Implementation Study. JMIR Res Protoc. 2020 Jul 14;9(7):e16319. doi: 10.2196/16319. PMID 32442144
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 11, 2019 and September 3, 2021, three-hundred forty-three (343) participants were approached for enrollment, two-hundred ninety-three (293) patients consented and were enrolled on study.
  Eighty nine (89) providers were recruited and gave verbal consent for participation.
Units Other Than Participants: SCDIC Study Sites
Groups:
- Sites 1, 2 (InCharge Health App) Sickle Cell Disease (SCD) Patients: Sites 1 and 2 Patients: Enrolled 11/11/2019 to 7/17/2020. Data collected 11/11/2019 to 7/17/2020, 7/17/2020 to 12/30/2020 post-intervention data collected .
  Patient received the InCharge Health app for 6 months. InCharge Health mobile application features include: Daily reminders; customizable messages; Symptom tracker; streaks; Graphing adherence against pain symptoms; communication features; and an education bank.
  Provider received the HU Toolbox app for 9 months HU Toolbox mobile application: The HU Toolbox app includes algorithms for hydroxyurea use. In addition, it has the NHLBI guidelines, and has the ability to search for key words, add notes, print PDF documents, and contact local SCD specialists.
- Sites 3, 4 (InCharge Health App) Sickle Cell Disease (SCD) Patients: Sites 3 and 4 Patients: Enrolled 6/11/2020 to 9/3/2021. Data collected 6/11/2020 to 9/3/2021 to 5/17/22 post-intervention data collected.
  Patient received the InCharge Health app for 6 months. InCharge Health mobile application features include: Daily reminders; customizable messages; Symptom tracker; streaks; Graphing adherence against pain symptoms; communication features; and an education bank.
  Provider received the HU Toolbox app for 9 months HU Toolbox mobile application: The HU Toolbox app includes algorithms for hydroxyurea use. In addition, it has the NHLBI guidelines, and has the ability to search for key words, add notes, print PDF documents, and contact local SCD specialists.
- Sites 5, 6, 7 (InCharge Health App) Sickle Cell Disease (SCD) Patients: Sites 5, 6 and 7 Patients: Enrolled 1/5/2021 to 9/3/2021. Data collected 1/5/2021 to 11/3/2021, 11/3/2021 to 7/7/2023 post-intervention data collected.
  Patient received the InCharge Health app for 6 months. InCharge Health mobile application features include: Daily reminders; customizable messages; Symptom tracker; streaks; Graphing adherence against pain symptoms; communication features; and an education bank.
  Provider received the HU Toolbox app for 9 months HU Toolbox mobile application: The HU Toolbox app includes algorithms for hydroxyurea use. In addition, it has the NHLBI guidelines, and has the ability to search for key words, add notes, print PDF documents, and contact local SCD specialists.
Period: Overall Study
Arm/Group | Sites 1, 2 (InCharge Health App) Sickle Cell Disease (SCD) Patients | Sites 3, 4 (InCharge Health App) Sickle Cell Disease (SCD) Patients | Sites 5, 6, 7 (InCharge Health App) Sickle Cell Disease (SCD) Patients
Started | 136; 2 SCDIC Study Sites | 99; 2 SCDIC Study Sites | 147; 3 SCDIC Study Sites
Patients-All Enrolled | 94; 2 SCDIC Study Sites | 88; 2 SCDIC Study Sites | 111; 3 SCDIC Study Sites
Providers-All Enrolled | 42; 2 SCDIC Study Sites | 11; 2 SCDIC Study Sites | 36; 3 SCDIC Study Sites
Patients-Completed | 84; 2 SCDIC Study Sites | 67; 2 SCDIC Study Sites | 110; 3 SCDIC Study Sites
Providers-Completed | 40; 2 SCDIC Study Sites | 9; 2 SCDIC Study Sites | 32; 3 SCDIC Study Sites
Completed | 124; 2 SCDIC Study Sites | 76; 2 SCDIC Study Sites | 142; 3 SCDIC Study Sites
Not Completed | 12; 0 SCDIC Study Sites | 23; 0 SCDIC Study Sites | 5; 0 SCDIC Study Sites
Not completed — Lost to Follow-up-Patients | 7 | 14 | 0
Not completed — Lost to Follow-up-Providers | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Withdrawal by Provider | 0 | 0 | 4
Not completed — Death-Patient | 2 | 1 | 0
Not completed — Hydroxyurea New Starts | 0 | 0 | 1
Not completed — Did not complete the baseline survey/activities | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients: Patient receives the InCharge Health app for 6 months
  InCharge Health mobile application: The InCharge Health app features include: Daily reminders; Ability to customize content of message and time of day when the message comes; Symptom tracker to monitor daily pain and mood; 7-day streak that tracks daily adherence; Graphing adherence against pain symptoms; Communication feature allowing the patient to connect to the clinic and a "health partner"; Link to discussion forum where communication to other patients can occur; Education bank that provides information about SCD and hydroxyurea. Participants can delay daily push notifications. If hospitalized, participants may stop notifications. A special feature of the app is to set up a "health partner", who may be a person the participant may choose from his/her contact list and who will receive notifications if it had been <4 hours since not documenting the use of hydroxyurea. The "app healthy partner" will be encouraged to message the participant to remind him/her to take the medication.
- Arm 2 (HU Toolbox App) - Providers: Provider receives the HU Toolbox app for 9 months
  HU Toolbox mobile application: The HU Toolbox app includes algorithms for hydroxyurea use and is ready for immediate use on Apple and Android operating systems. In addition, it has the NHLBI guidelines adapted for pediatrics (guidelines/recommendations separated by age) and for adults (guidelines/ recommendations separated by organ system, laboratory, or physical exam finding). The HU Toolbox app includes the ability to search guidelines for key words and add notes. Algorithms are also included as PDF documents that can be printed out or emailed. Finally, a contact list of local SCD specialists and important contacts is included, so providers can easily contact SCD experts and expect an answer in 24 hours or less. The HU Toolbox app is easily updated with all data and resources stored on a cloud-based server that can provide instant up-to-date information to those using the app.
- Total: Total of all reporting groups
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients | Arm 2 (HU Toolbox App) - Providers | Total
Number analyzed (Participants) | 293 | 89 | 382
Age, Customized [Count of Participants; unit: Participants]
  15-17 years | 23 | 0 | 23
  18-24 years | 97 | 0 | 97
  25-44 years | 168 | 53 | 221
  45-64 years | 5 | 28 | 33
  65 years and older | 0 | 5 | 5
  Unknown | 0 | 3 | 3
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 151 | 65 | 216
  Male | 141 | 20 | 161
  Unknown | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 84 | 95
  Not Hispanic or Latino | 279 | 3 | 282
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 1 | 16 | 17
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 283 | 24 | 307
  White | 2 | 47 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Sickle cell disease genotype (n, %) [Count of Participants; unit: Participants] — Population: Data for Sickle cell disease genotype collected for patient participants only.
  Participants
    number analyzed (Participants) | 293 | 0 | 293
    HbSS/HbSβ0-thalassemia | 246 | 0 | 246
    HbSC/HbSβ+- thalassemia/other | 46 | 0 | 46
    Missing | 1 |  | 1
Marital Status [Count of Participants; unit: Participants] — Population: Data for Marital Status collected for patient participants only.
  Participants
    number analyzed (Participants) | 293 | 0 | 293
    Married/living as married | 30 | 0 | 30
    Never married | 242 | 0 | 242
    Divorced/separated/widowed | 11 | 0 | 11
    Missing | 10 | 0 | 10
Education (n, %) [Count of Participants; unit: Participants] — Population: Data for Education collected for patient participants only.
  Participants
    number analyzed (Participants) | 293 | 0 | 293
    Less than high school/Some high school | 43 |  | 43
    High school graduate or some college/vocational training | 176 |  | 176
    College Graduate+ | 66 |  | 66
    Missing | 8 |  | 8
Employment [Count of Participants; unit: Participants] — Population: Data for Employment collected for patient participants only.
  Participants
    number analyzed (Participants) | 293 | 0 | 293
    Employed | 95 | 0 | 95
    Not employed by choice (homemaker, student, retired) | 75 | 0 | 75
    Not employed, other (laid off/sick leave/maternity leave, unemployed, disabled) | 115 | 0 | 115
    Missing | 8 | 0 | 8
Annual Income (n, %) [Count of Participants; unit: Participants] — Population: Data for Annual Income collected for patient participants only.
  Participants
    number analyzed (Participants) | 293 | 0 | 293
    $25,000 or less | 166 |  | 166
    $25,001-$50,000 | 60 |  | 60
    $50,001-$100,000+ | 40 |  | 40
    Missing | 27 |  | 27
Provider Type, n (%) [Count of Participants; unit: Participants] — Population: Data for Provider Type collected for providers only.
  Participants
    number analyzed (Participants) | 0 | 89 | 89
    Physician |  | 49 | 49
    Nurse Practitioner or Physician Assistant |  | 36 | 36
    Chose not to report |  | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in PDC From Baseline Through 24 Weeks
Description: The primary outcome is the change in the percentage of days covered (PDC) of hydroxyurea, measured by comparing PDC during the 24-week baseline interval (i.e. prior the intervention) with PDC during the 24-week follow-up interval. PDC is calculated as the number of days covered (i.e., days of prescription refill dates and supply of each prescription) divided by the number of days in a treatment time point then multiply by 100 to obtain the PDC as a percentage.
Time Frame: baseline (prior to the intervention), week 24
Population: Of the 293 patients enrolled, 235 patients were analyzed. 21 were lost to follow-up, 13 were missing 24-week refill data, 12 had incomplete baseline refill data, 5 were new hydroxyurea starts, 3 involuntarily discontinued hydroxyurea, 2 died, and 2 were withdrawn from the study.
Measure: Mean (Standard Deviation); unit: percentage of days
Groups:
- Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients: Sickle cell patients meeting the eligibility requirements for the study.
  Patient receives the InCharge Health app for 6 months
  InCharge Health mobile application: The InCharge Health app features include: Daily reminders; Ability to customize content of message and time of day when the message comes; Symptom tracker to monitor daily pain and mood; 7-day streak that tracks daily adherence; Graphing adherence against pain symptoms; Communication feature allowing the patient to connect to the clinic and a "health partner"; Link to discussion forum where communication to other patients can occur; Education bank that provides information about SCD and hydroxyurea. Participants can delay daily push notifications. If hospitalized, participants may stop notifications. A special feature of the app is to set up a "health partner", who may be a person the participant may choose from his/her contact list and who will receive notifications if it had been <4 hours since not documenting the use of hydroxyurea. The "app healthy partner" will be encouraged to message the participant to remind him/her to take the medication.
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 235
percentage of days | 16.3 (33.1)

2. Secondary Outcome: Implementation of InCharge Health App.
Description: Count of all enrolled patients who used the InCharge Health app at least once during the study period among all enrolled
Time Frame: baseline, 24 weeks
Population: 293 participants data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients: Sickle cell patients who used the InCharge Health app at least once during the study period.
  InCharge Health mobile application: The InCharge Health app was used for 6 months. Its features include: Daily reminders; Ability to customize content of message and time of day when the message comes; Symptom tracker to monitor daily pain and mood; 7-day streak that tracks daily adherence; Graphing adherence against pain symptoms; Communication feature allowing the patient to connect to the clinic and a "health partner"; Link to discussion forum where communication to other patients can occur; Education bank that provides information about SCD and hydroxyurea. Participants can delay daily push notifications. If hospitalized, participants may stop notifications. A special feature of the app is to set up a "health partner", who may be a person the participant may choose from his/her contact list and who will receive notifications if it had been <4 hours since not documenting the use of hydroxyurea. The "app healthy partner" will be encouraged to message the participant to remind him/her to take the medication.
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 293
Participants | 240

3. Secondary Outcome: Change in Mean Corpuscular Volume (MCV)
Description: Mean difference between MCV during the baseline interval and during the follow-up interval
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the outcome analysis, 228 patients were analyzed for this outcome as 7 had missing data
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 228
fL | 0.70 (0.50)

4. Secondary Outcome: Change in Fetal Hemoglobin
Description: Mean difference between fetal hemoglobin during the baseline interval and during the follow-up interval
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the outcome analysis, 137 patients were analyzed for this outcome as 98 had missing data
Measure: Mean (Standard Deviation); unit: percentage of Hemoglobin F
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 137
percentage of Hemoglobin F | 1.78 (0.76)

5. Secondary Outcome: Change in Hemoglobin Concentration
Description: Mean difference between hemoglobin during the baseline interval and during the follow-up interval
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the outcome analysis, 228 patients were analyzed for this outcome as 7 had missing data
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 228
g/dL | 0.05 (0.07)

6. Secondary Outcome: Change in Reticulocyte Percentage
Description: Mean difference between reticulocyte percentage during the baseline interval and during the follow-up interval
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the outcome analysis, 193 patients were analyzed for this outcome as 42 had missing data
Measure: Mean (Standard Deviation); unit: percentage of reticulocytes
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 193
percentage of reticulocytes | -1.48 (0.49)

7. Secondary Outcome: Change in Absolute Neutrophil Percentage
Description: Mean difference between neutrophil percentage during the baseline interval and during the follow-up interval
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the primary outcome analysis, 198 patients were analyzed for this outcome as 37 had missing data
Measure: Mean (Standard Deviation); unit: percentage of neutrophils
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 198
percentage of neutrophils | 0.93 (1.01)

8. Secondary Outcome: Change Bilirubin
Description: Mean difference between total bilirubin during the baseline interval and during the follow-up interval
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the primary outcome analysis, 214 patients were analyzed for this outcome as 21 had missing data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 214
mg/dL | -0.09 (0.10)

9. Secondary Outcome: Change in Mean Plasma Lactate Dehydrogenase (LDH)
Description: Mean difference between LDH during the baseline interval and during the follow-up interval
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the primary outcome analysis, 101 patients were analyzed for this outcome as 134 had missing data
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 101
IU/L | -18.8 (18.5)

10. Secondary Outcome: Change in Rate of Emergency Room Visits Per Patient in the Last 24 Weeks
Description: Mean difference between number of emergency room visits during the baseline interval and during the follow-up interval.
Time Frame: baseline, 24 weeks
Population: Of the 293 patients enrolled, 235 patients were analyzed for this outcome as 58 did not complete the 24 weeks
Measure: Mean (Standard Deviation); unit: emergency room visits per patient
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 235
emergency room visits per patient | 0.35 (1.94)

11. Secondary Outcome: Change in Rate of Hospitalization Per Patient in the Last 24 Weeks
Description: Mean difference between number of hospitalizations during the baseline interval and during the follow-up interval.
Time Frame: baseline, 24 weeks
Population: Of the 293 patients enrolled, 235 patients were analyzed for this outcome as 58 did not complete the 24 weeks
Measure: Mean (Standard Deviation); unit: Number of hospitalizations per patients
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 235
Number of hospitalizations per patients | 0.01 (0.84)

12. Secondary Outcome: Change in Patient Reported Pain Quality
Description: Mean difference between scores on the Patient Reported Outcomes Information System (PROMIS) Pain Quality Scale during baseline and follow-up when the responses, never, rarely, sometimes, often, and always are coded 0 through 4. The Patient Reported Outcomes Information System (PROMIS) Pain Quality Scale has a minimum value of "never", coded as 0, and a maximum value of "always", coded as 4 for analysis. A higher score indicates worse pain.
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the primary outcome analysis, 182 patients were analyzed for this outcome as 53 had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 182
score on a scale | 0.15 (0.15)

13. Secondary Outcome: Change in Patient Reported Pain Impact: ASCQ-Me Pain Impact Scale
Description: Mean difference between scores on the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Pain Episode Frequency and Severity Scale during baseline and follow-up when the responses, never, rarely, sometimes, often, and always are coded 0 through 4. Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Pain Episode Frequency and Severity Scale has a minimum value of "never", coded as 0, and a maximum value of "always", coded as 4 for analysis. A higher score indicates worse pain.
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the primary outcome analysis, 187 patients were analyzed for this outcome as 48 had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 187
score on a scale | -0.005 (1.090)

14. Secondary Outcome: Change in Patient Reported Pain Frequency and Severity
Description: as for outcome 13
Time Frame: baseline, 24 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 187
score on a scale | 0 (1.24)

15. Secondary Outcome: Change in Healthy Literacy
Description: Mean difference between responses to the Single item literacy screener (SILS) during baseline and follow-up when the responses, Never, rarely, sometimes, often, and always are coded 0 through 4; score is the sum of responses to 8 questions (score range: 0-32). The Single item literacy screener (SILS) has a minimum value of "never", coded as 0, and a maximum value of "always", coded as 4 for analysis. A higher score means lower health literacy.
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the primary outcome analysis, 183 patients were analyzed for this outcome as 52 had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 183
score on a scale | 0.05 (1.00)

16. Secondary Outcome: Change in Perceived Self-efficacy
Description: Mean difference between responses to the Patient reported outcomes information system (PROMIS) medication self-efficacy short form during baseline and follow-up when the responses, I am not at all confident, I am a little confident, I am somewhat confident, I am quite confident, and I am very confident are coded 0 to 4. The Patient Reported Outcomes Information System (PROMIS) Pain Quality Scale has a minimum value of "I am not at all confident", coded as 0, and a maximum value of "I am very confident", coded as 4 for analysis. A higher score indicates greater self-efficacy.
Time Frame: baseline, 24 weeks
Population: Of the 235 patients included in the primary outcome analysis, 232 patients were analyzed for this outcome as 2 had missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 232
score on a scale | -3.9 (12.8)

17. Secondary Outcome: Change in Provider Knowledge of Hydroxyurea (HU) Prescription Guidelines
Description: Mean difference between responses during baseline and follow-up to the 5 questions on the Hydroxyurea Knowledge Scale regarding knowledge of correctly prescribing hydroxyurea. Each question was scored 0 (incorrect response) or 1 (correct) and the 5 scores were summed to produce totals of 0 to 5.
Time Frame: baseline, 9 months
Population: 69 of 89 providers analyzed because of missing data
Measure: Mean (Standard Deviation); unit: number of correctly answered questions
Groups:
- Arm 2 (HU Toolbox App) - Providers: Physicians and advanced level practitioners meeting the eligibility requirements for the study.
  HU Toolbox mobile application: The HU Toolbox app includes algorithms for hydroxyurea use and is ready for immediate use on Apple and Android operating systems. In addition, it has the NHLBI guidelines adapted for pediatrics (guidelines/recommendations separated by age) and for adults (guidelines/ recommendations separated by organ system, laboratory, or physical exam finding). The HU Toolbox app includes the ability to search guidelines for key words and add notes. Algorithms are also included as PDF documents that can be printed out or emailed. Finally, a contact list of local SCD specialists and important contacts is included, so providers can easily contact SCD experts and expect an answer in 24 hours or less. The HU Toolbox app is easily updated with all data and resources stored on a cloud-based server that can provide instant up-to-date information to those using the app.
Arm/Group | Arm 2 (HU Toolbox App) - Providers
Number analyzed (Participants) | 69
number of correctly answered questions | 0.14 (0.71)

18. Secondary Outcome: Change is Provider Self-efficacy of Hydroxyurea (HU) Prescription Guidelines
Description: Hydroxyurea self-efficacy scale (comfort level and perceived effectiveness in prescribing hydroxyurea) with responses scored 0 to 4. The Hydroxyurea self-efficacy scale has a minimum value of "very uncomfortable", coded as 0 and a maximum value of "very comfortable", coded as 4. A higher score indicates greater self-efficacy.
Time Frame: baseline, 9 months
Population: 69 of 89 providers analyzed because of missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 2 (HU Toolbox App) - Providers
Number analyzed (Participants) | 69
score on a scale | 0.07 (1.71)

19. Secondary Outcome: Mean Change in PDC From Baseline Through 36 Weeks
Description: This outcome is the change in the percentage of days covered (PDC) of hydroxyurea, measured by comparing PDC during the 24-week baseline interval (i.e. prior the intervention) with PDC during the 36-week follow-up interval. PDC is calculated as the number of days covered (i.e., days of prescription refill dates and supply of each prescription) divided by the number of days in a treatment time point then multiply by 100 to obtain the PDC as a percentage.
Time Frame: baseline (prior to the intervention), week 36
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percentage of days covered
Groups:
- Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients: Sickle cell patients meeting the eligibility requirements for the study.
  InCharge Health mobile application: The InCharge Health app features include: Daily reminders; Ability to customize content of message and time of day when the message comes; Symptom tracker to monitor daily pain and mood; 7-day streak that tracks daily adherence; Graphing adherence against pain symptoms; Communication feature allowing the patient to connect to the clinic and a "health partner"; Link to discussion forum where communication to other patients can occur; Education bank that provides information about SCD and hydroxyurea. Participants can delay daily push notifications. If hospitalized, participants may stop notifications. A special feature of the app is to set up a "health partner", who may be a person the participant may choose from his/her contact list and who will receive notifications if it had been <4 hours since not documenting the use of hydroxyurea. The "app healthy partner" will be encouraged to message the participant to remind him/her to take the medication.
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
Number analyzed (Participants) | 232
percentage of days covered | 11.75 (33.65)

ADVERSE EVENTS:
Time Frame: Patient participants were followed for adverse events from baseline to 24 weeks.
Arm/Group | Arm 1 (InCharge Health App) - Sickle Cell Disease (SCD) Patients
All-Cause Mortality (participants affected / at risk) | 3/293
Serious Adverse Events (participants affected / at risk) | 0/293
Other Adverse Events (participants affected / at risk) | 0/293

LIMITATIONS AND CAVEATS:
Due to the onset of the Covid 1-19 pandemic and delays with the IRB at several institutions, we had to move to a staggered enrollment instead of a full stepped wedge design. The process was outlined in the paper under Citations.

The Covid-19 pandemic also caused clinic lockdowns which impacted the implementation of the mHealth intervention at some sites. Sites were able to adapt recruitment and implementation measures to continue the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT04080167/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT04080167/ICF_000.pdf